CLINICAL TRIAL: NCT04601233
Title: Testosterone TReatment for Erectile Dysfunction in Male Multiple Sclerosis Patients With Low Testosterone (TTRED-MS Study)
Brief Title: Testosterone Treatment for Erectile Dysfunction and Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1288
Record Dates: First submitted 2020-10-02; First posted 2020-10-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Erectile Dysfunction; Testosterone Deficiency
Keywords: Multiple Sclerosis; Erectile Dysfunction; Testosterone Deficiency
MeSH Terms: conditions — Multiple Sclerosis; Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Single open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment open label arm (Experimental): Open-label feasibility study to determine the effects of testosterone (Xyosted 75mg subcutaneous once per week for 3 months) on erectile function in male Multiple Sclerosis patients with low testosterone.
  Interventions: Drug: XYOSTED 75 milligram (mg) in 0.5 ML Auto-Injector

INTERVENTIONS:
Drug: XYOSTED 75 milligram (mg) in 0.5 ML Auto-Injector — Self injection testosterone treatment

SUMMARY:
The purpose of the study is to determine the effects of testosterone treatment on erectile function, fatigue, depression, cognitive function, quality of life, urinary incontinence, pain, and damage to neurons in male Multiple Sclerosis patients with low testosterone, using questionnaires, blood samples and a rectal exam in volunteers 55 years and older.

DETAILED DESCRIPTION:
Volunteers will be treated weekly with Xyosted 75 mg (given subcutaneously) for 3 months during which they will have 3 study visits, 6 weeks apart. The Baseline visit will include providing a blood sample, completing questionnaires, receiving training on the Xyosted auto-injector, and undergoing a rectal exam for participants 55 years and older. Visits 2 and 3 will also include collecting a blood sample and completing questionnaires. At Visit 3, the rectal exam for those age 55 years and older will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 18 years and older, with a definite diagnosis of multiple sclerosis.
* Low testosterone (<300 ng/dl) on two successive blood draws before 9:00 am
* Not in an intercurrent relapse.
* Sexually active.
* Have subjective complaints about erectile function and libido.
* Must be willing and able to get labs drawn, complete questionnaires (BDI, MFIS, MSNQ, SDMT, MSQOL, ADAM, AUASS, SHIM, MSHQ, ICIQ, UDI, IIQ, MPQ) and commit to site visits schedule.

Exclusion Criteria:

* Males unable to fulfill the above criteria and all female patients.
* Males who have been on sex hormone treatment including androgens, estrogens, or anti-estrogens for hypogonadism or other medical condition during the 12 months prior to study.
* Males who have taken dehydroepiandrosterone (DHEA) during the 3 months prior to study.
* Patients who are taking anticoagulants or have thrombosis, serious cardiac, pulmonary, renal, gastrointestinal, hepatic, immunologic, infectious, neoplastic (with particular focus on patients with known or suspected estrogen or testosterone-dependent tumors), urologic disease especially prostatic hypertrophy/nodules and testicular mass, or insulin-dependent diabetes.
* Patients with an abnormal prostate as evidenced by known history of prostatic disease, symptoms suggestive of prostatic disease or elevated levels of prostatic specific antigen (PSA 4 ng/ml or higher) measured within the last 12 months.
* Patients with history or complaint of testicular mass.
* Patients with hematocrit greater than 50%
* Patients with major psychiatric illness
* Patients with active alcoholism.
* Patients with a history of drug abuse within the past five years.
* Patients with BMI ≥ 35
* Patients with generalized skin disease that may affect absorption of testosterone (e.g. psoriasis) or a known skin intolerance to alcohol.
* Patients with history of pituitary disease.
* Patients with a cholesterol level greater than 300 mg/dl.
* Patients who are receiving or have received experimental therapies in the six months preceding enrollment.
* Patients who have history of positive titers to Human Immunodeficiency Virus (HIV)1 and 2; HTLV1; or Venereal Disease Research Laboratory (VDRL).
* Patients who have clinical evidence of Lyme disease.
* Males who are trying to get their partner pregnant.
* Patients on Finasteride
* Patients who are mentally or emotionally incompetent in the opinion of the examining neurologist or unable to give informed consent, or to understand and comply with the study protocol.
* Any other contraindications according to the manufacturer's exclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the change in self-reported erectile function from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using Androgen Deficiency in the Aging Male (ADAM score). | Change from baseline to 12 weeks
  Androgen Deficiency in the Aging Male (ADAM score) includes ten "Yes or No" questions, with an answer "Yes" to number 1 or 7 or if you answer "Yes" to more than 3 questions, you may have low Testosterone.
Determine the change in self-reported erectile function from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using Sexual Health in Men (SHIM score). | Change from baseline to 12 weeks
  Sexual Health in Men (SHIM score) with a range of 1 to 25 with a higher number representing less erectile dysfunction.
Determine the change in self-reported erectile function from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using Male Sexual Health Questionnaire short form (MSHQ-SF). | Change from baseline to 12 weeks
  Male Sexual Health Questionnaire short form (MSHQ-SF) with a range of 1 to 15 with a higher number representing better ejaculatory function, in addition to one bother/satisfaction question, scored 1 to 5 where the higher represents more bothersome.

SECONDARY OUTCOMES:
Measure the change in self-reported fatigue from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the Modified Fatigue Impact Scale (MFIS). | Change from baseline to 12 weeks
  Modified Fatigue Impact Scale (MFIS) with a range of 0 to 84 with a higher number representing greater impact of fatigue on a person's activities.
Measure the change in self-reported depression from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the Beck Depression Inventory (BDI). | Change from baseline to 12 weeks
  Beck Depression Inventory (BDI) with a range of 0 to 63 with a higher number representing higher level of depression.
Measure the change in cognitive function from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the Symbol Digit Modalities Test (SDMT). | Change from baseline to 12 weeks
  Symbol Digit Modalities Test (SDMT) which provides a score for as many items as can be completed in 90 seconds (t-score calculated using age, sex and education normative data), with a higher score representing a better performance.
Measure the change in cognitive function from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the Multiple Sclerosis Neuropsychological Screening Questionnaire (MSNQ). | Change from baseline to 12 weeks
  Multiple Sclerosis Neuropsychological Screening Questionnaire (MSNQ) with a range of 0 to 30 with a higher number representing worse cognitive function.
Measure the change in self-reported overall quality of life from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the Multiple Sclerosis Quality of Life Scale (MSQOL-54). | Change from baseline to 12 weeks
  Multiple Sclerosis Quality of Life Scale (MSQOL-54) which goes from 0 to 100 with a higher score indicating a better quality of life.
Measure the change in self-reported urinary incontinence from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the American Urological Association Symptom Score (AUASS). | Change from baseline to 12 weeks
  The American Urological Association Symptom Score (AUASS) with a range of 0 to 35 with a higher number representing more severe enlarged prostate symptoms.
Measure the change in self-reported urinary incontinence after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using International Consultation on Incontinence Questionnaire short form (ICIQ-SF). | Change from baseline to 12 weeks
  International Consultation on Incontinence Questionnaire short form (ICIQ-SF) with a range of 0 to 21 with a higher number representing greater impairment from incontinence.
Measure the change in self-reported urinary incontinence from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using Urogenital Distress Inventory short form (UDI-6). | Change from baseline to 12 weeks
  Urogenital Distress Inventory short form (UDI-6) with a range of 0 to 100 with a higher number representing higher the disability.
Measure the change in self-reported urinary incontinence from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using Incontinence Impact Questionnaire short form (IIQ-7). | Change from baseline to 12 weeks
  Incontinence Impact Questionnaire short form (IIQ-7) with a range of 0 to 100 with a higher number representing greater impact by urinary incontinence on the person's life.
Measure the change in self-reported pain from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the McGill Pain Questionnaire (MPQ). | Change from baseline to 12 weeks
  McGill Pain Questionnaire (MPQ) with a range of 0 to 78 with a higher number representing greater pain.
Measure the change in Multiple Sclerosis lesions, indirectly from baseline to 12-weeks after 12 weeks of treatment with XYOSTED in males with Multiple Sclerosis with low testosterone using the serum levels of neurofilament-light chains (NF-L). | Change from baseline to 12 weeks
  The serum levels of neurofilament-light chains (NF-L) with a higher level representing more neuro-axonal injury in the central nervous system.

CONTACTS AND LOCATIONS:
Overall Officials: Omar A Raheem, MD, Principal Investigator — Assistant Professor, Urology
Locations (1):
- LSU Health Multispecilaity Clinics, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bove R, Musallam A, Healy BC, Raghavan K, Glanz BI, Bakshi R, Weiner H, De Jager PL, Miller KK, Chitnis T. Low testosterone is associated with disability in men with multiple sclerosis. Mult Scler. 2014 Oct;20(12):1584-92. doi: 10.1177/1352458514527864. Epub 2014 Apr 7. PMID 24710799
- [Background] Tehranipour M, Moghimi A. Neuroprotective effects of testosterone on regenerating spinal cord motoneurons in rats. J Mot Behav. 2010 May-Jun;42(3):151-5. doi: 10.1080/00222891003697921. PMID 20363715
- [Background] Sicotte NL, Giesser BS, Tandon V, Klutch R, Steiner B, Drain AE, Shattuck DW, Hull L, Wang HJ, Elashoff RM, Swerdloff RS, Voskuhl RR. Testosterone treatment in multiple sclerosis: a pilot study. Arch Neurol. 2007 May;64(5):683-8. doi: 10.1001/archneur.64.5.683. PMID 17502467
- [Background] Young CA, Tennant A; TONiC Study Group. Sexual functioning in multiple sclerosis: Relationships with depression, fatigue and physical function. Mult Scler. 2017 Aug 1;23(9):1268-1275. doi: 10.1177/1352458516675749. Epub 2016 Nov 1. PMID 28681643
- [Background] Cunningham GR, Stephens-Shields AJ, Rosen RC, Wang C, Bhasin S, Matsumoto AM, Parsons JK, Gill TM, Molitch ME, Farrar JT, Cella D, Barrett-Connor E, Cauley JA, Cifelli D, Crandall JP, Ensrud KE, Gallagher L, Zeldow B, Lewis CE, Pahor M, Swerdloff RS, Hou X, Anton S, Basaria S, Diem SJ, Tabatabaie V, Ellenberg SS, Snyder PJ. Testosterone Treatment and Sexual Function in Older Men With Low Testosterone Levels. J Clin Endocrinol Metab. 2016 Aug;101(8):3096-104. doi: 10.1210/jc.2016-1645. Epub 2016 Jun 29. PMID 27355400
- [Background] Yassin AA, Saad F. Treatment of sexual dysfunction of hypogonadal patients with long-acting testosterone undecanoate (Nebido). World J Urol. 2006 Dec;24(6):639-44. doi: 10.1007/s00345-006-0120-0. PMID 17048032